CLINICAL TRIAL: NCT05538130
Title: A PHASE 1A/B OPEN-LABEL MASTER STUDY OF PF-07799544 AS A SINGLE-AGENT AND IN COMBINATION WITH OTHER TARGETED AGENTS IN PARTICIPANTS WITH BRAF-MUTANT MELANOMA AND OTHER SOLID TUMORS
Brief Title: A Study to Learn About the Study Medicine Called PF-07799544 as Monotherapy or in Combination in People With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4901001; NCT05538130 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Melanoma; Glioma; Thyroid Cancer; Non-Small Cell Lung Cancer; Malignant Neoplasms; Brain Neoplasms; Advanced or Metastatic Solid Tumors; HGG; LGG; Low Grade Glioma; High Grade Glioma; Differentiated Thyroid Cancer; NSCLC (Non-small Cell Lung Cancer)
Keywords: solid tumors; BRAF; advanced solid tumors; B-Raf; MAPK; neoplasms; BRAF V600
MeSH Terms: conditions — Melanoma; Glioma; Thyroid Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a Monotherapy Dose Escalation (Experimental): Participants will receive PF-07799544
  Interventions: Drug: PF-07799544
- Phase 1b Combination Dose Escalation (Experimental): Participants will receive PF-07799544 and PF-07799933
  Interventions: Drug: PF-07799544; Drug: PF-07799933
- Phase 1b Combination Dose Expansion (Experimental): Participants will receive PF-07799544 and PF-07799933
  Interventions: Drug: PF-07799544; Drug: PF-07799933

INTERVENTIONS:
Drug: PF-07799544 — Tablet
  Other Names: ARRY-134
Drug: PF-07799933 — Tablet
  Other Names: ARRY-440
  Arms: Phase 1b Combination Dose Escalation; Phase 1b Combination Dose Expansion

SUMMARY:
The purpose of this clinical trial is to learn the safety and effects of the study medicine (PF-07799544) alone or in combination as a potential cancer treatment for adults with advanced solid tumors. The study will be conducted in two parts: PF-07799544 as a single agent (Phase 1a) and PF-07799544 in combination with another study medicine called PF-07799933 (Phase 1b).

Phase 1a is no longer open for enrollment. In Phase1b (noted as "this study"), we are seeking participants who have:

* a solid tumor which is metastatic or recurrent (excluding colorectal cancer)
* tumor with the mutation (abnormal gene) called "BRAF V600"
* received required prior treatment for cancer per cohort assigned.

All participants in this study will receive both study medicines. Both study medicines are tablets that are taken by mouth at home twice a day.

Participants will receive study medicines until their cancer is no longer responding, unacceptable side effects, or 2 years. Participants may continue to receive study therapy beyond 2 years. We will examine the experiences of people receiving the study medicines. This will help us determine if the study medicines are safe and effective.

ELIGIBILITY:
Phase 1b Inclusion Criteria:

* Diagnosis of advanced/metastatic solid tumor (excluding colorectal cancer)
* Measurable disease by RECIST version 1.1
* Evidence of a BRAF V600 mutation
* Prior therapy per tumor cohort
* Adequate organ function per protocol

Phase 1b Exclusion Criteria:

* Other active malignancy within 3 years
* Presence of leptomeningeal disease
* History or current evidence of retinal vein occlusion (RVO) or history of retinal degenerative disease
* Concurrent neuromuscular disorder associated with elevated creatine kinase (CK)
* Active gastrointestinal disease as defined per protocol
* History of interstitial lung disease as defined per protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2027-04-08 (Estimated); Study Completion 2028-10-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1a monotherapy and Phase 1b combination dose escalation: Number of participants with dose limiting toxicities (DLTs) | Cycle 1 (21 days)
  DLTs will be evaluated during the first cycle (21 days) as a single agent (phase 1a monotherapy) or in combination with other agents (phase 1b dose escalation)
Phase 1a monotherapy and Phase 1b combination dose escalation: Number of participants with treatment-emergent adverse events (AEs) | Baseline to 28 days after last dose of study medication
  AEs as characterized by type, frequency, severity, timing, seriousness, and relationship to study therapy
Phase 1a monotherapy and Phase 1b combination dose escalation: Number of participants with clinically significant change from baseline in laboratory abnormalities | Baseline to 28 days after last dose of study treatment
  Laboratory abnormalities as characterized by type, frequency, severity, and timing.
Phase 1a monotherapy and Phase 1b combination dose escalation: Number of participants with clinically significant change from baseline in vital sign abnormalities | Baseline to 28 days after last dose of study treatment
  Vital sign abnormalities as characterized by type, frequency, severity, and timing.
Phase 1a monotherapy and Phase 1b combination dose escalation: Number of participants with clinically significant change from baseline in physical exam abnormalities | Baseline to 28 days after last dose of study treatment
  Physical exam abnormalities as as graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Phase 1b Dose Expansion: Overall response rate (ORR) | Baseline to 2 years
  Response will be evaluated via radiographical tumor assessments by RECIST v1.1 for solid tumors or RANO for primary brain tumors

SECONDARY OUTCOMES:
Phase 1a monotherapy and Phase 1b combination dose escalation: ORR | Baseline to 2 years
  ORR as assessed using the RECIST version 1.1.
Phase 1b Dose Expansion: Number of participants with treatment-emergent adverse events (AEs) | Baseline to 2 years
  AEs as characterized by type, frequency, severity, timing, seriousness, and relationship to study therapy
Phase 1b Dose Expansion: Number of participants with clinically significant change from baseline in vital sign abnormalities | Baseline to 2 years
  Vital sign abnormalities as characterized by type, frequency, severity, and timing.
Phase 1b Dose Expansion: Number of participants with clinically significant change from baseline in laboratory abnormalities | Baseline to 2 years
  Laboratory abnormalities as characterized by type, frequency, severity, and timing.
Phase 1b Dose Expansion: Duration of Response (Overall and in CNS) | Baseline to 2 years
  Response will be evaluated via radiographical tumor assessments by RECIST v1.1 for solid tumors or RANO for primary brain tumors
Phase 1b Dose Expansion: Intracranial response | Baseline to 2 years
  Intracranial response by RECIST version 1.1 (for brain metastases)
Phase 1b Dose Expansion: Progression Free Survival (PFS) | Baseline to 2 years
  Response will be evaluated via radiographical tumor assessments by RECIST v1.1 for solid tumors or RANO for primary brain tumors
PK Parameters: Maximum Observed Concentration (Cmax) | Baseline to 2 years
  Single dose and multiple dose PK will be calculated as data permits
PK Parameters: Maximum Plasma Concentration (Tmax) | Baseline to 2 years
  Single dose and multiple dose PK will be calculated as data permits
PK Parameters: Area Under Curve (AUC) | Baseline to 2 years
  Single dose and multiple dose PK will be calculated as data permits
PK Parameters: terminal elimination half-life (t½) | Baseline to 2 years
  Singe dose and multiple dose PK will be calculated as data permits
PK Parameters: Apparent Oral Clearance (CL/F) | Baseline to 2 years
  Singe dose and multiple dose PK will be calculated as data permits
PK Parameters: Apparent Volume of Distribution (Vz/F) | Baseline to 2 years
  Singe dose and multiple dose PK will be calculated as data permits

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (75):
- United States (56):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham - Phase I Clinical Trials Unit, Birmingham, Alabama
  - Highlands Oncology Group, PA, Fayetteville, Arkansas
  - Highlands Oncology Group, PA, Rogers, Arkansas
  - Highlands Oncology Group, PA, Springdale, Arkansas
  - The Angeles Clinic and Research Institute- A Cedars-Sinai Affiliate, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCSF Medical Center, Investigational Pharmacy, San Francisco, California
  - The Angeles Clinic and Research Institue, A Cedars-Sinai Affiliate (Emergency Back-up only), Santa Monica, California
  - Moffitt Cancer Center, Richard M. Shulze Family Foundation Outpatient Center, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt McKinley Hospital, Tampa, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigitte Harris Cancer Pavilion, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - HealthPartners Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Methodist Hospital Inpatient Pharmacy, Saint Louis Park, Minnesota
  - HealthPartners Cancer Center at regions Hospital, Saint Paul, Minnesota
  - Regions Hospital Pharmacy, Saint Paul, Minnesota
  - MSK Basking Ridge., Basking Ridge, New Jersey
  - MSK Monmouth., Middletown, New Jersey
  - MSK Bergen., Montvale, New Jersey
  - Optum Medical Care, PC, Brewster, New York
  - MSK Commack., Commack, New York
  - MSK Westchester., Harrison, New York
  - Laura & Isaac Perlmutter Cancer Center - NYU ACC, New York, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - NYU Langone Faculty Group Practice, New York, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - Memorial Sloan Kettering Cancer Center 53rd street., New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Columbia University Medical Center - Neurological Institute of New York, New York, New York
  - CUIMC Research Pharmacy, New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - Brooklyn Radiation Oncology, PC, Richmond Hill, New York
  - MSK Nassau., Uniondale, New York
  - Clinical Research Alliance, Westbury, New York
  - Cleveland Clinic Taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute- Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Australia (3):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Brazil (3):
  - ANIMI - Unidade de Tratamento Oncologico, Lages, Santa Catarina
  - Centro de Oncologia - CEON+ - Unidade São Caetano do Sul, São Caetano do Sul, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino, São Paulo
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus, Québec, Quebec
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China
- Israel (5):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Soroka Medical Center, Beersheba, Southern District
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4901001